CLINICAL TRIAL: NCT03482895
Title: Endocrine and Absorptive Intestinal Function in Patients at Two Years of Bariatric Surgery: Omega Loop Gastric Bypass Versus Roux-en-Y Gastric Bypass
Brief Title: MINI Bypass Versus Roux-en-Y Bypass: Differences in HOrmonal Secretions at 2 Years of Surgery
Acronym: MINIBHO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société Francophone Nutrition Clinique et Métabolisme (Other)
Responsible Party: Sponsor
Other Study IDs: K171007J; 2017-A02816-47 (Other: France: ANSM)
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Bariatric Surgery
Keywords: Gastric Bypass; Intestinal Absorption; Gastrointestinal Hormones; Enteroendocrine Cells
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Blood sampling & Feces sampling: Blood samplings at different times after a meal test: 0, 15, 30, 60, 90 and 120 minutes.
  Feces sampling: collection during 24 hours
  Interventions: Biological: Blood sampling; Biological: Feces sampling

INTERVENTIONS:
Biological: Blood sampling — Quantitative analysis of enterohormones, citrulline and ApoB48
Biological: Feces sampling — Intestinal absorption assessment

SUMMARY:
Gastric bypass with omega loop technic (OLGB) seems to be as effective as gastric bypass roux-en-Y (RYGB the reference) for the management of obesity and type 2 diabetes, but with less early surgical complications and more undernutrition in long terms.

This study aims to explore the profile of secretion of entero-insular hormone after a meal test in OLGB patient vs RYGB to understand the mechanisms of the improvement of type 2 diabetes after OLGB.

Secondary objectives are to better understand the absorptive function of the gut after a gastric bypass, to understand why is there more undernutrition in long term after OLGB than after RYGB.

DETAILED DESCRIPTION:
In the treatment of obesity associated with type 2 diabetes, there is still few informations comparing the gastric bypass roux-en-Y (RYGB), the reference method, and the bypass in Omega (OLGB). The effectiveness of both interventions is comparable regarding weight loss and the management of type 2 diabetes but the level of proof remains low. Nutritional deficiencies and chronic diarrhea are reported in both interventions. It seems that the OLGB would cause more malabsorption and undernutrition but the OLGB would lead to less early operative complications because it has only one gastro-jejunal anastomosis compared to RYGB which has two.

The success of the RYGB for the remission of diabetes, is partly associated with a change in secretion's profile of intestinal hormones participating in the glucose homeostasis, especially the GLP-1. There is no studies published reporting the level of secretion (fasting or postprandial) of gastrointestinal hormones after OLGB. It is important to understand how this surgery produces its effects, especially on diabetes.

MINIBHO main hypothesis is that the secretion's profile of entero-insular hormones, like GLP-1, are exacerbated after OLGB just like in RYGB, that would explain the same level of improvement of T2 diabetes after both surgery.

Kinetic study of entero-insular secretion will be assessed by some blood dosages of entero-insular hormones (GLP-1, GLP-2, Gastric inhibitory polypeptide (GIP), glicentine, Insulin, peptide C, Glucagon and glucose) in 30 patients (15 OLGB and 15 RYGB). These dosages will be made at different times after a meal test (during fasting, 15 minutes, 30 minutes, 60 minutes, 90 minutes and 120 minutes after the meal) to search a significant difference in the profile of secretion between the OLGB and RYGB patients.

Investigators also hypothesize that the editing method of the OLGB leads to a decrease in the food absorption profile compared to RYGB. To explore this hypothesis, citrulline and apolipoprotein B48 (ApoB48) levels will be measured, which reflect enterocyte function of the patients, and will be compared between patients operated with RYGB vs OLGB. Functional enterocyte mass will be correlated to the absorptive function of the gut which will be evaluated by the examination of the 24h feces.

The main objective is to determine whether the secretion profiles of entero-insular hormone during a meal are different or not in patients operated with OLGB compared to RYGB. The secondary objectives are to evaluate in these patients the absorptive function and the functional enterocyte mass.

ELIGIBILITY:
Inclusion Criteria:

* Roux en Y gastric bypass or omega loop gastric bypass at two years of the surgery (6 months more or less)
* 18 years minimum
* weight > 40kg

Exclusion Criteria:

* Type 1 diabetes diagnosed with the positivity of anti Glutamate Acid Decarboxylase (GAD) or anti Ia2
* Treatment with Insulin, Glucagon Like Peptide 1 (GLP1) or anti-DiPeptidyl Peptidase-4 (DPP4) during the study
* Unbalanced type 2 diabetes : HbA1c > 8%
* Anemia with hemoglobin < 7g/dl
* Gut inflammatory disease ; infectious disease, cancer, iatrogenic disease, auto-immune disease
* Pregnant or breastfeeding women
* allergy to Carmin (E120)
* participation to another clinical trial
* patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient recruited 2 years (+/- 6 months) after Omega-loop Gastric Bypass or Roux-en-Y Gastric Bypass
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Kinetic of GLP-1 secretion | 0, 15, 30, 60, 90 and 120 minutes after a meal test
  Area under the plasma concentration versus time curve of GLP-1

SECONDARY OUTCOMES:
Plasmatic dosage of citrulline | Baseline
  Plasmatic concentration of Citrulline versus enterocyte mass function
Plasmatic dosage of Apolipoprotein B48 | Baseline
  Plasmatic concentration of Apolipoprotein B48 versus enterocyte mass function
Lipidic Absorptive Coefficient | 1 day
  Percentage between lipidic food intakes and lipidic excretion in feces
Protein Absorptive Coefficient | 1 day
  Percentage between protein food intakes and protein excretion in feces
Glucidic Absorptive Coefficient | 1 day
  Percentage between carbohydrate food intakes and carbohydrate excretion in feces
kinetic of GLP-2 secretion | 0, 15, 30, 60, 90 and 120 minutes after a meal test
  Area under the plasma concentration versus time curve of GLP-2
Kinetic of GIP secretion | 0, 15, 30, 60, 90 and 120 minutes after a meal test
  Area under the plasma concentration versus time curve of GIP
Kinetic of Peptide C secretion | 0, 15, 30, 60, 90 and 120 minutes after a meal test
  Area under the plasma concentration versus time curve of Peptide C
Kinetic of Insulin secretion | 0, 15, 30, 60, 90 and 120 minutes after a meal test
  Area under the plasma concentration versus time curve of Insulin
Kinetic of Glucagon secretion | 0, 15, 30, 60, 90 and 120 minutes after a meal test
  Area under the plasma concentration versus time curve of Glucagon
Kinetic of Glicentin secretion | 0, 15, 30, 60, 90 and 120 minutes after a meal test
  Area under the plasma concentration versus time curve of Glicentin
Kinetic of Glycemia | 0, 15, 30, 60, 90 and 120 minutes after a meal test
  Area under the plasma concentration versus time curve of glucose

CONTACTS AND LOCATIONS:
Overall Officials: Claire Carette, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP - Hôpital Européen Georges-Pompidou, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Bandt D, Rives-Lange C, Frigout Y, Bergerot D, Blanchard A, Le Gall M, Lacorte JM, Chevallier JM, Czernichow S, Poghosyan T, Carette C, Le Beyec J. Similar Gut Hormone Secretions Two Years After One Anastomosis Gastric Bypass and Roux-en-Y Gastric Bypass: a Pilot Study. Obes Surg. 2022 Mar;32(3):757-762. doi: 10.1007/s11695-021-05837-5. Epub 2022 Jan 7. PMID 34993850